CLINICAL TRIAL: NCT03953924
Title: Effects of Transtheoretical Model-based Intervention and Motivational Interviewing on the Management of Depression in Hospitalized Patients With Coronary Heart Disease : A Randomized, Controlled Trial
Brief Title: TTM-based Intervention and MI in CHD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, SiLan Yang, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SYang
Record Dates: First submitted 2019-05-11; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Coronary Heart Disease; Depression
Keywords: transtheoretical model; motivational interviewing; depression; coronary heart disease
MeSH Terms: conditions — Coronary Disease; Depression | interventions — Methods; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: No interventions were performed for the control patients during study. However, they received conventional care (Simple and unstructured patient education about diet, exercise and so on).
  Patients in the intervention group received conventional care, TTM-based intervention and MI. The intervention was provided by nurses who were trained, including two researchers and a general nurse of cardiovascular ward. The primary researcher was leader of the study. The leader explained the purpose, significance and methods of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The leader of this study entered the cardiovascular medical ward and screened potential eligible patients according to medical records in each hospital. Leaders informed the purpose, significance, methods, sessions of the study to patients. Patients were randomly divided into two groups by using a block randomization list with a block size of 4 at 1:1. A research assistant put the generated random number into opaque consecutively numbered envelopes and sealed the envelopes, and then handed it to enrolling researchers. When enrolling a new participant, the enrolling investigators opened the sealed envelope after participant's name was written on next available envelopes. A sequentially numbered and opaque, sealed envelope system was used by a non-investigator. Additionally, all data collection was conducted by another research assistant who was blind to the study design and allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No interventions were performed for the control patients during the study. While those in the control group were given conventional care ( nursing procedure, education about diet, exercise and so on)
- Intervention group (Experimental): The patients in intervention group received conventional care, transtheoretical model-based (TTM-based) intervention and motivational interviewing (MI).
  Interventions: Other: Transtheoretical model-based (TTM - based) intervention and motivational interviewing (MI)

INTERVENTIONS:
Other: Transtheoretical model-based (TTM - based) intervention and motivational interviewing (MI) — The MI was implemented 2 times, 20 minutes each time, the trained nurse interviewed each patient face-to-face by bedside. Based on the evaluation results and motivational interviewing, the change stages of the patients' behavior changes were identified. According to the changing stage,TTM - based intervention was given 3 times in the form of a small course, 20 minutes each time, the key point was divided into three stages.
  Arms: Intervention group

SUMMARY:
In the middle of this century, coronary heart disease (CHD) is the most common cause of death in the United States. Chinese health service survey showed that about 1000,0000 ~ 320,000 people were suffering from CHD in the mainland of China in 2008. The high mortality and morbidity of CHD will aggravate the psychological burden of patients, such as depression. Depression is the most psychological problem in CHD patients. The incidence of depression in Chinese population was in the range of 4%~6%, while it was as high as 14%~17% in patients with CHD. Depression not only affects the patients' illness, but also reducing their quality of life, the compliance of drugs and lifestyle. In addition, depression is a major risk factor for the mortality and morbidity of cardiovascular disease. Therefore, it's urgently needed to screen and treat the depression of patients with CHD.

At present, the treatment of depression in patients with CHD mainly includes antidepressant, cognitive behavioral therapy， psychological counseling, knowledge education, relaxation therapy and so on. However, the medicine would yield side - effect. Furthermore, the content of psychological interventions are not systematic and dynamic. Moreover, patients' depressive level varies in different periods, the traditional psychological intervention just focused on the ultimate psychological benefits, and cannot analyze some factors and staged results in the process of psycho-behavioral change. Thus, an dynamic and effective intervention to alleviate depression in patients with CHD is imperative.

DETAILED DESCRIPTION:
The transtheoretical model (TTM) is a purposeful behavioral change model. It is a systematic study of people's behavior change based on a variety of theories. Effective outcomes with TTM also have been applied in many studies of health behavior change, especially in the field of two aspects: on the one hand, to change unhealthy behaviors such as smoking, drinking, weight control and so on. Besides, a way to involve individuals in health behavior change is motivational interviewing (MI). MI is a way that taking patients as the center approach to interpersonal communication, which helps patients discover and overcome their ambivalence, thereby triggering behavioral changes. A study showed that MI might have favorable effects on changing patients' depression and found that the effect of a single use of MI was better than that of cognitive-behavioral therapy. In summary, the TTM-based interventions and MI were used to change behavior fields. To our knowledge, few studies have been conducted to determine the effects of the TTM-based intervention and MI on depression. Therefore, this study decided to determine the effects of TTM-based intervention and MI on the management of depression in hospitalized patients with CHD.

The aim of this study was to determine the effects of TTM-based intervention and MI on patients' stages of change, processes of change, decisional balance, self-efficacy, and depression. The study's hypothesis was: (1) The patients in the intervention group would be a positive shift in stages of change, the scores of cognitive level, behavioral level, perceived benefits, self-efficacy, perceived barriers and depression after intervention compared with the control group.

The sample comprised 110 (each group: 55) patients with coronary heart disease (CHD) in the Medicine-Cardiovascular Departments of three hospitals in Changsha.

The whole trail was on the basis of the CONSORT statements and a single, blind, randomized, controlled trial. Study procedures were approved by the institutional review boards of all participating All patients were recruited by enrolling researchers for eligibility and then enrolled in the study if they were eligible and informed consent. Patients were randomly divided into two groups by using a block randomization list with a block size of 4 at 1:1.

A research assistant put the generated random number into opaque consecutively numbered envelopes and sealed the envelopes, and then handed it to enrolling researchers. When the eligible patients were recruited in the study, the enrolling researchers numbered the patients, opening the same numbers sealed envelopes. The enrolling researchers were blind about the design of this study.

The patients in the intervention group received conventional care, TTM-based intervention and MI; Interventions were provided by trained nurses. First, The leader of this research contacted the hospital, getting the consent of the relevant departments and ward heads of the hospital to screen research objects before the beginning of the study, telling patients the purpose, significance, methods of the research, times to fill out the questionnaire, and the possible risks and benefits of the study.

The MI was implemented 2 times, 20 minutes each time, the trained nurses interviewed each patient face-to-face in the unit. Data were collected at 2 time points: the patient was on admission (T, obtain the baseline information) and the patient was 2- days before discharged (T0, obtain the information after intervention), according to the assessment of their current stage of change and depression delivered by filling the Stages of Change Subscale and Hamilton Rating Scale. TTM - based intervention was given 3 times in the form of a small course, 20 minutes each time according to the changing stage.

No interventions were performed for the control group participants during the study. However, these patients received conventional care ( nursing procedure, education about diet, exercise and so on).

Data were collected by a research assistant who was blind to the study design and allocation of participants. At baseline, sociodemographic and clinical characteristics were collected from medical records and personal interviews.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Be diagnosed as coronary heart disease (typical clinical angina manifestations, electrocardiogram changes, and coronary angiography) confirmed by the World Health Organization / International Cardiology in October 1997 and cardiac function is graded from I to III;
* Must be volunteered to participate in the study;
* Must be conscious with clear communication ability.

Exclusion Criteria:

* Had cerebrovascular accident, malignant tumor, malignant hypertension(systolic pressure >180 and/or diastolic pressure >100 mmHg);
* Had a psychiatric history or serious cognitive conscious obstacles;
* Had been participated in other similar research subjects;
* No mobile phone or home phone is available for contacts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Stage of change for coronary heart disease patients with depression | 2 - days (T0) before discharge.
  The subscale was used for measuring the stages of individual depression management behavior, it consisted of one item and five statements(precontemplation, contemplation, preparation, action, maintenance). The scale has good reliability and the retest reliability and the reliability was 0.790.
Process of change for coronary heart disease patients with depression | 2 - days (T0) before discharge.
  Process of change subscale was used to evaluated individuals' experiences or activities that can influence individuals to take effective measures to manage depression. It had 30 items. Each item was scored from 1 (never) to 5 (always). The higher the dimension score, the higher the frequency of use of the process. The Cronbach's alpha of experimental processes and behavioral processes was 0.786, 0.817.
Decisional balance for coronary heart disease patients with depression | 2 - days (T0) before discharge.
  The subscale was used to assess the importance of individuals to take effective methods to manage depression and determine the importance of taking action. It comprised 12 items and two dimensions that perceived benefits and perceived barriers. Each item was scored from 1 (not important) to 5 (extremely important). The Cronbach's alpha of perceived benefits and perceived barriers was 0.690, 0.700.
Self-efficacy for coronary heart disease patients with depression: scale | 2 - days (T0) before discharge.
  The subscale consisted of 6 items. Each item was scored from 1 (no confidence at all) to 5 (full of confidence), the scores reflect the degree of confidence in managing depression effectively. Higher scores reflect higher confidence. The Cronbach's alpha of subscale was 0.735.
Hamilton Rating Scale for Depression | 2 - days (T0) before discharge.
  The scale was compiled in 1960 by Hamilton, including 24 items. A few items (4th, 5th, 6th, 12tn, 14th, 16th, 17th, 18th, 21st items) were evaluated with 0-2 points scoring method, the rest of the items were divided into 0-4 points scoring method. Higher total scores reflect serious depression. In this study, Cronbach's alpha was 0.819.

SECONDARY OUTCOMES:
Social Demographic Data Recording Form | on admission (T).
  Patients' demographic information was obtained from the social demographic data recording form and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Zhang, PhD., Study Chair — Central South University

IPD SHARING:
Plan to Share IPD: No
The process of data collection cost a lot of human and material resources,some of the data was privacy information of participants, and so on.Considering this, it is improper to share these data.

REFERENCES:
- [Result] Aghaei M, Samkhaniyan E, Mahdavi A, Faraji J, Roshandel Z. Effectiveness of behavioral-cognitive group therapy on depression, anxiety, and stress of patients with coronary heart disease. J Med Life. 2015;8(Spec Iss 4):252-257. PMID 28316740
- [Result] Albus C, Ladwig KH, Herrmann-Lingen C. [Psychocardiology: clinically relevant recommendations regarding selected cardiovascular diseases]. Dtsch Med Wochenschr. 2014 Mar;139(12):596-601. doi: 10.1055/s-0033-1360102. Epub 2014 Mar 11. German. PMID 24619718
- [Result] Anastopoulou K, Fradelos EC, Misouridou E, Kourakos M, Berk A, Papathanasiou IV, Kleisiaris C, Zyga S. Moderating Nutritious Habits in Psychiatric Patients Using Transtheoretical Model of Change and Counseling. Adv Exp Med Biol. 2017;988:63-71. doi: 10.1007/978-3-319-56246-9_5. PMID 28971389
- [Result] Arri SS, Ryan M, Redwood SR, Marber MS. Mental stress-induced myocardial ischaemia. Heart. 2016 Mar;102(6):472-80. doi: 10.1136/heartjnl-2014-307306. Epub 2016 Jan 4. No abstract available. PMID 26729692
- [Result] Belialov FI. [Depression, anxiety, and stress in patients with coronary heart disease]. Ter Arkh. 2017;89(8):104-109. doi: 10.17116/terarkh2017898104-109. Russian. PMID 28914859
- [Result] Blumenthal JA, Babyak MA, O'Connor C, Keteyian S, Landzberg J, Howlett J, Kraus W, Gottlieb S, Blackburn G, Swank A, Whellan DJ. Effects of exercise training on depressive symptoms in patients with chronic heart failure: the HF-ACTION randomized trial. JAMA. 2012 Aug 1;308(5):465-74. doi: 10.1001/jama.2012.8720. PMID 22851113
- [Result] Alcantara C, Muntner P, Edmondson D, Safford MM, Redmond N, Colantonio LD, Davidson KW. Perfect storm: concurrent stress and depressive symptoms increase risk of myocardial infarction or death. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):146-54. doi: 10.1161/CIRCOUTCOMES.114.001180. Epub 2015 Mar 10. PMID 25759443
- [Result] Carney RM, Freedland KE. Depression and coronary heart disease. Nat Rev Cardiol. 2017 Mar;14(3):145-155. doi: 10.1038/nrcardio.2016.181. Epub 2016 Nov 17. PMID 27853162
- [Result] Dalen JE, Alpert JS, Goldberg RJ, Weinstein RS. The epidemic of the 20(th) century: coronary heart disease. Am J Med. 2014 Sep;127(9):807-12. doi: 10.1016/j.amjmed.2014.04.015. Epub 2014 May 5. PMID 24811552
- [Result] Skaal L, Pengpid S. The predictive validity and effects of using the transtheoretical model to increase the physical activity of healthcare workers in a public hospital in South Africa. Transl Behav Med. 2012 Dec;2(4):384-391. doi: 10.1007/s13142-012-0136-5. Epub 2012 May 31. PMID 23293685
- [Result] Evers KE, Prochaska JO, Johnson JL, Mauriello LM, Padula JA, Prochaska JM. A randomized clinical trial of a population- and transtheoretical model-based stress-management intervention. Health Psychol. 2006 Jul;25(4):521-9. doi: 10.1037/0278-6133.25.4.521. PMID 16846327
- [Result] Hammadah M, Al Mheid I, Wilmot K, Ramadan R, Shah AJ, Sun Y, Pearce B, Garcia EV, Kutner M, Bremner JD, Esteves F, Raggi P, Sheps DS, Vaccarino V, Quyyumi AA. The Mental Stress Ischemia Prognosis Study: Objectives, Study Design, and Prevalence of Inducible Ischemia. Psychosom Med. 2017 Apr;79(3):311-317. doi: 10.1097/PSY.0000000000000442. PMID 28002382
- [Result] Hoy J, Natarajan A, Petra MM. Motivational Interviewing and the Transtheoretical Model of Change: Under-Explored Resources for Suicide Intervention. Community Ment Health J. 2016 Jul;52(5):559-67. doi: 10.1007/s10597-016-9997-2. Epub 2016 Feb 17. PMID 26886871
- [Result] Johnson SS, Paiva AL, Cummins CO, Johnson JL, Dyment SJ, Wright JA, Prochaska JO, Prochaska JM, Sherman K. Transtheoretical model-based multiple behavior intervention for weight management: effectiveness on a population basis. Prev Med. 2008 Mar;46(3):238-46. doi: 10.1016/j.ypmed.2007.09.010. Epub 2007 Oct 23. PMID 18055007
- [Result] Lange-Asschenfeldt C, Lederbogen F. [Antidepressant therapy in coronary artery disease]. Nervenarzt. 2011 May;82(5):657-64; quiz 665-6. doi: 10.1007/s00115-010-3181-7. German. PMID 21109992
- [Result] Lee WW, Choi KC, Yum RW, Yu DS, Chair SY. Effectiveness of motivational interviewing on lifestyle modification and health outcomes of clients at risk or diagnosed with cardiovascular diseases: A systematic review. Int J Nurs Stud. 2016 Jan;53:331-41. doi: 10.1016/j.ijnurstu.2015.09.010. Epub 2015 Oct 3. PMID 26493130
- [Result] Lee YM, Park NH, Kim YH. Process of change, decisional balance, self-efficacy and depression across the stages of change for exercise among middle aged women in Korea. Taehan Kanho Hakhoe Chi. 2006 Jun;36(4):587-95. doi: 10.4040/jkan.2006.36.4.587. PMID 16825842
- [Result] Levesque DA, Van Marter DF, Schneider RJ, Bauer MR, Goldberg DN, Prochaska JO, Prochaska JM. Randomized trial of a computer-tailored intervention for patients with depression. Am J Health Promot. 2011 Nov-Dec;26(2):77-89. doi: 10.4278/ajhp.090123-QUAN-27. PMID 22040388
- [Result] Lichtman JH, Bigger JT Jr, Blumenthal JA, Frasure-Smith N, Kaufmann PG, Lesperance F, Mark DB, Sheps DS, Taylor CB, Froelicher ES; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Epidemiology and Prevention; American Heart Association Interdisciplinary Council on Quality of Care and Outcomes Research; American Psychiatric Association. Depression and coronary heart disease: recommendations for screening, referral, and treatment: a science advisory from the American Heart Association Prevention Committee of the Council on Cardiovascular Nursing, Council on Clinical Cardiology, Council on Epidemiology and Prevention, and Interdisciplinary Council on Quality of Care and Outcomes Research: endorsed by the American Psychiatric Association. Circulation. 2008 Oct 21;118(17):1768-75. doi: 10.1161/CIRCULATIONAHA.108.190769. Epub 2008 Sep 29. PMID 18824640
- [Result] Lim SH, Chan SW, He HG. Patients' Experiences of Performing Self-care of Stomas in the Initial Postoperative Period. Cancer Nurs. 2015 May-Jun;38(3):185-93. doi: 10.1097/NCC.0000000000000158. PMID 24836957
- [Result] Lippke S, Schwarzer R, Ziegelmann JP, Scholz U, Schuz B. Testing stage-specific effects of a stage-matched intervention: a randomized controlled trial targeting physical exercise and its predictors. Health Educ Behav. 2010 Aug;37(4):533-46. doi: 10.1177/1090198109359386. Epub 2010 Jun 14. PMID 20547760
- [Result] Marcus BH, Bock BC, Pinto BM, Forsyth LH, Roberts MB, Traficante RM. Efficacy of an individualized, motivationally-tailored physical activity intervention. Ann Behav Med. 1998 Summer;20(3):174-80. doi: 10.1007/BF02884958. PMID 9989324
- [Result] Orth-Gomer K, Schneiderman N, Wang HX, Walldin C, Blom M, Jernberg T. Stress reduction prolongs life in women with coronary disease: the Stockholm Women's Intervention Trial for Coronary Heart Disease (SWITCHD). Circ Cardiovasc Qual Outcomes. 2009 Jan;2(1):25-32. doi: 10.1161/CIRCOUTCOMES.108.812859. Epub 2009 Jan 6. PMID 20031809
- [Result] Pajak A, Jankowski P, Kotseva K, Heidrich J, de Smedt D, De Bacquer D; EUROASPIRE Study Group. Depression, anxiety, and risk factor control in patients after hospitalization for coronary heart disease: the EUROASPIRE III Study. Eur J Prev Cardiol. 2013 Apr;20(2):331-40. doi: 10.1177/2047487312441724. Epub 2012 Mar 6. PMID 22396247
- [Result] Pizzi C, Costa GM, Santarella L, Flacco ME, Capasso L, Bert F, Manzoli L. Depression symptoms and the progression of carotid intima-media thickness: a 5-year follow-up study. Atherosclerosis. 2014 Apr;233(2):530-536. doi: 10.1016/j.atherosclerosis.2014.01.012. Epub 2014 Jan 21. PMID 24530790
- [Result] Prochaska JO, Butterworth S, Redding CA, Burden V, Perrin N, Leo M, Flaherty-Robb M, Prochaska JM. Initial efficacy of MI, TTM tailoring and HRI's with multiple behaviors for employee health promotion. Prev Med. 2008 Mar;46(3):226-31. doi: 10.1016/j.ypmed.2007.11.007. Epub 2007 Nov 22. PMID 18155287
- [Result] Prochaska JO, Velicer WF, Rossi JS, Goldstein MG, Marcus BH, Rakowski W, Fiore C, Harlow LL, Redding CA, Rosenbloom D, et al. Stages of change and decisional balance for 12 problem behaviors. Health Psychol. 1994 Jan;13(1):39-46. doi: 10.1037//0278-6133.13.1.39. PMID 8168470
- [Result] Prochaska JO, Velicer WF, Fava JL, Rossi JS, Tsoh JY. Evaluating a population-based recruitment approach and a stage-based expert system intervention for smoking cessation. Addict Behav. 2001 Jul-Aug;26(4):583-602. doi: 10.1016/s0306-4603(00)00151-9. PMID 11456079
- [Result] Miller WR, Rollnick S. Meeting in the middle: motivational interviewing and self-determination theory. Int J Behav Nutr Phys Act. 2012 Mar 2;9:25. doi: 10.1186/1479-5868-9-25. No abstract available. PMID 22385872
- [Result] Rubak S, Sandbaek A, Lauritzen T, Christensen B. Motivational interviewing: a systematic review and meta-analysis. Br J Gen Pract. 2005 Apr;55(513):305-12. PMID 15826439
- [Result] Summers KM, Martin KE, Watson K. Impact and clinical management of depression in patients with coronary artery disease. Pharmacotherapy. 2010 Mar;30(3):304-22. doi: 10.1592/phco.30.3.304. PMID 20180613
- [Result] Velicer WF, Prochaska JO. An expert system intervention for smoking cessation. Patient Educ Couns. 1999 Feb;36(2):119-29. doi: 10.1016/s0738-3991(98)00129-3. PMID 10223017
- [Result] Zhu LX, Ho SC, Sit JW, He HG. The effects of a transtheoretical model-based exercise stage-matched intervention on exercise behavior in patients with coronary heart disease: a randomized controlled trial. Patient Educ Couns. 2014 Jun;95(3):384-92. doi: 10.1016/j.pec.2014.03.013. Epub 2014 Mar 29. PMID 24726785 (Retraction: PMID 24976395 J Adv Nurs. 2014 Oct;70(10):2414)
- [Derived] Li X, Yang S, Wang Y, Yang B, Zhang J. Effects of a transtheoretical model - based intervention and motivational interviewing on the management of depression in hospitalized patients with coronary heart disease: a randomized controlled trial. BMC Public Health. 2020 Mar 30;20(1):420. doi: 10.1186/s12889-020-08568-x. PMID 32228532